CLINICAL TRIAL: NCT02018757
Title: Clinical Application Study of Transarterial Chemoembolization Containing Arsenic Trioxide in the Treatment of Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Arsenic Trioxide Contained in TACE in the Treatment of HCC
Acronym: SEATH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Hospital of China Medical University (Other)
Collaborators: Sun Yat-sen University (Other); Zhongda Hospital (Other); Fudan University (Other); Xijing Hospital (Other)
Responsible Party: Principal Investigator, Haibo Shao, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012AA022701
Record Dates: First submitted 2013-12-09; First posted 2013-12-23 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular; primary liver cancer; primary hepatocellular carcinoma; transarterial chemoembolization; Chemoembolization, Therapeutic; arsenic trioxide; arsenous anhydride; diarsenic trioxide; randomized controlled trial; multicenter study; HCC; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- As2O3 (Experimental): Subjects will be treated with TACE containing As2O3
  Interventions: Drug: TACE containing As2O3
- placebo (Placebo Comparator): Subjects will be treated with TACE containing placebo which mimics the arsenic trioxide
  Interventions: Drug: TACE containing placebo

INTERVENTIONS:
Drug: TACE containing As2O3 — transarterial chemoembolization containing a mixture of 20mg of arsenic trioxide, 40mg of adriamycin and some dose of 40% ultra-fluid lipiodol
  Other Names: transarterial chemoembolization,TACE,As2O3,arsenious acid
  Arms: As2O3
Drug: TACE containing placebo — transarterial chemoembolization containing a mixture of 20mg of placebo, 40mg of adriamycin and some dose of 40% ultra-fluid lipiodol
  Arms: placebo

SUMMARY:
The purpose of the study is to determine whether transarterial chemoembolization containing arsenic trioxide is safe and effective in the treatment of intermediate-stage hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* accordance with primary hepatocellular carcinoma diagnosis standard：cytohistology standard or non-invasive standard.1）+2）a or 1）+2）b+3）of the following are the non-invasive diagnosis criteria:(1)patients with HBV or HCV related liver cirrhosis.(2)radiological lesion(s) in liver with arterial hypervascularity and venous or delayed phase washout: a.one kind of imaging technology diagnosis for those with lesions>2cm;b.two kinds of imaging technology obtains the consistent conclusion for lesions with diameter of 1-2 cm.(3)serum AFP level ≥400 ug/L lasting for more than 1 month or ≥200 ug/L lasting for more than 2 months, other diseases that may cause the AFP level increase can be excluded,such as pregnancy, genital or embryonic tumors and active hepatitis.
* age of 18 to 75 year,male or female
* life expectancy of 12 weeks
* Barcelona Clinic Liver Cancer (BCLC)stage B
* laboratory tests:(1)leukocyte>3*19^9/L;(2)hemoglobin≥8.5g/dl;(3)platelet count ≥50*10^9/L,(4)ALT and AST were less than three times the normal limit;(5)albumin ≥ 3.0 g/dl;(6)total bilirubin acuities 3 mg/dl;(7)prothrombin time international standardization ratio (PT - INR) < = 2.3 or prothrombin time (PT)more than normal compared 3 seconds;(8)serum creatinine is less than 1.5 times the normal of the upper limit
* patients with signed informed consent

Exclusion Criteria:

* concomitant malignancies distinct from HCC currently or previously
* allergic to subject agent(such as arsenic) or other agent related to the trial
* BCLC stage 0,A,C or D
* HCC accounting for the 70% of the liver size or more
* liver function Child-Pugh score of C
* ECOG score of 1 or higher
* severe heart diseases,such as congestive heart failure with cardiac function of New York Heart Association(NYHA)functional class II or severe, active coronary disease(except for who with myocardial infarction for more than 6 months) and cardiac arrhythmia needing medical management(except for that controllable by β-blockers、calcium channel blockers and digoxin )
* uncontrollable hypertension(diastolic blood pressure cannot be controlled below 90 mmHg even after antihypertension treatment by antihypertensive drugs).
* active severe infection(grade 2 or higher according to NCI-CTCAE version 4.0)
* active tuberculosis or pulmonary tuberculosis cannot be excluded
* CNS malignancies, including intracranial metastases
* gastrointestinal bleeding with clinical findings in the previous 30 days
* chronic renal failure
* pregnancy or breastfeeding
* any other unstable conditions or circumstances possibly to jeopardise the safety or compliance of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
time to progression | From date of randomization until the date of first documented progression, up to 24 months

SECONDARY OUTCOMES:
objective response rate | every 3 months from randomization until the date of first documented progression, up to 24 months
  patients proportion of CR and PR according to mRECIST
progression free survival | From date of randomization until the date of first documented progression, up to 24 months
  survival from randomization to the date of first documented progression according to the mRECIST criterion
overall survival | From date of randomization until the date of death from any cause, up to 60 months
Proportion of Participants with Adverse Events | every 3 months from randomization until the date of first documented progression, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Shao, MD,PhD, Principal Investigator — First Hospital of China Medical University
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Xijing Hospital，Fourth Military Medical University, Xi'an, Shaanxi
  - Zhongshan Hospital Fudan University, Shanghai